CLINICAL TRIAL: NCT00617318
Title: Pomegranate Products for Prevention of Common Cold and Influenza-Like Symptoms: A Double- Blind, Placebo-Controlled Randomized Clinical Trial
Brief Title: Pomegranate Products for Prevention of Common Cold
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Texas Heart Institute (Other)
Collaborators: POM Wonderful LLC (Industry)
Responsible Party: Mohammad Madjid, Texas Heart Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: POM001
Record Dates: First submitted 2008-02-06; First posted 2008-02-18 (Estimated); Last update posted 2008-02-18 (Estimated); Status verified 2007-11

CONDITIONS: Influenza; Common Cold; Cough; Headache; Fever
Keywords: Pomegranate; Influenza; Common Cold; Cough; Severity; Efficacy
MeSH Terms: conditions — Influenza, Human; Common Cold; Cough; Headache; Fever

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental)
  Interventions: Dietary Supplement: Pomegranate
- B (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Pomegranate — All subjects were randomized and assigned to a 16-week treatment with either POM concentrate or placebo. The placebo matched the taste, smell, and appearance of the POM concentrate. Supplies were shipped to the investigation site in equal proportions marked as "A" and "B," and site personnel did not know the code. The treatment products (POM concentrate or placebo) were supplied as 2-oz packages, each containing a single day's consumption, and were dispensed as packages of 33 units (a 4-week plus 5-day supply). The subjects were to consume one 2 oz. package daily for a period of 16 weeks.
  Arms: A
Dietary Supplement: Placebo — All subjects were randomized and assigned to a 16-week treatment with either POM concentrate or placebo. The placebo matched the taste, smell, and appearance of the POM concentrate. Supplies were shipped to the investigation site in equal proportions marked as "A" and "B," and site personnel did not know the code. The treatment products (POM concentrate or placebo) were supplied as 2-oz packages, each containing a single day's consumption, and were dispensed as packages of 33 units (a 4-week plus 5-day supply). The subjects were to consume one 2 oz. package daily for a period of 16 weeks.
  Arms: B

SUMMARY:
Pomegranate has a long history of use in folk medicine. There is vast data on the health benefits of pomegranate fruit and juice. Multiple studies have established the strong antioxidative effects of pomegranate polyphenols (primarily the ellagitannin punicalagin) and their health effects. A vast number of animal and human clinical studies have provided evidence on effect of pomegranate products on improving blood lipid profile, reducing blood pressure, improving endothelial function, anti-tumor activity, and its anti-atherosclerotic activity. We studied the protective effect of a pomegranate concentrate (POM Flu and Cold Formula®) in decreasing the incidence and duration of influenza-like illnesses and common cold among healthy adults.

DETAILED DESCRIPTION:
Pomegranate has a long history of use in folk medicine. Widely grown and consumed in most countries, pomegranate fruit and its products are now being produced and used more extensively in the US. The health benefits of pomegranate fruit and juice have been substantiated by much research, including multiple studies that have shown the beneficial antioxidative effects of pomegranate polyphenols (primarily ellagitannin punicalagin). Both in vitro and in vivo studies have demonstrated that pomegranate products provide hepatoprotection against toxins, reduce tumor cell growth, and have anti-angiogenesis, immunomodulatory, and free-radical scavenging effects. Furthermore, both animal and clinical studies indicate that pomegranate products can improve the blood lipid profile, reduce blood pressure, enhance endothelial function, and provide anti-tumor and anti-atherosclerotic activities.

No adverse events have been reported in clinical studies of more than 300 human subjects who consumed 8 fluid ounces (oz) or more of POM Wonderful® (POM LLC, Los Angeles, CA) pomegranate juice daily for periods as long as 3 years. These clinical trials have included sensitive subpopulations, such as patients with atherosclerotic disease, diabetes, hypertension, or prostate cancer. Moreover, no serious adverse effects have been reported in human, animal and in vitro studies published to date.

Ex vivo laboratory studies have shown that pomegranate polyphenols have considerable antioxidant activity. Because of the importance of oxidative stress in influenza infection and its complications, we previously assessed the anti-influenza effects of pomegranate products in ex vivo studies (See accompanying manuscript). Our laboratory findings showing the anti-influenza, virucidal effects of pomegranate products led us to study their clinical effects against influenza and the common cold in human volunteers. Previous studies have shown the effects of natural products on the incidence and course of influenza infection.

The purpose of the current study was to assess the effect of a pomegranate concentrate (POM Flu and Cold Formula, POM Wonderful LLC, Los Angeles, CA) in preventing the symptoms of influenza and common cold during the influenza season. POM Flu and Cold Formula is intended for oral use to provide supplemental antioxidants to a healthy population.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the inclusion criteria in order to be eligible to participate in the study:

* Subject must be able to read and sign Informed Consent Form (ICF).
* Subject must be male or female > 21 and < 49 years of age at the time the ICF is signed.
* Subject must have made a personal decision NOT to receive influenza vaccine this season.

Exclusion Criteria:

A subject meeting any of the exclusion criteria at baseline will be excluded from study participation:

* Subject who has a known allergy to pomegranate and POM products. Subject who has an intercurrent infection and fever during the week before the investigational product administration is to begin.

Subject who has experienced acute respiratory tract infection, otitis media, bronchitis or sinusitis, or who had been treated with an antiviral drug, systemic steroids, or immunosuppressants within two weeks of the Screening/Randomization Visit.

Subject who has uncontrolled chronic medical disorders (e.g., subjects with evidence of evolving hepatic or renal failure, congestive heart failure Killip Class IV, or any terminal disease).

* Subject who reports HIV infection.
* Subject who abuses alcohol or other drugs of abuse.
* Subject who has clinical evidence of current malignancy.
* Female subject with positive pregnancy test, or who is sexually active and not using adequate contraception regularly, or who is a nursing mother.
* Subject who has taken other experimental products within one month prior to study entry.
* Subject who has any medical condition that may interfere with study protocol adherence.
* Subject has any disorder (excluding illiteracy or visual impairment) that compromises the ability of the subject to give written informed consent and/or to comply with study procedures.
* Subject who in the opinion of the study investigator has a risk of non-compliance with study procedures, or cannot read, understand or complete study related materials.
* Subject who has a foreseeable inability to complete the scheduled follow-ups.
* Subject who meets one or more of the criteria for influenza immunization according to the current CDC List of Priority Groups for Vaccination.

Ages: 21 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 461 (Actual)
Dates: Start 2007-01; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure will be the incidence and severity of common cold using the modified severity scoring system during the sixteen week period of the POM Flu and Cold Formula use. | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Madjid, MD, Principal Investigator — Texas Heart Institute
Locations (1):
- Site 01, San Diego, California, United States